CLINICAL TRIAL: NCT00951288
Title: Effect of Saffron Supplementation on Macular Cone-mediated Function in Age-related Macular Degeneration
Acronym: safAMD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Benedetto Falsini, Associate Professor, Ophthalmology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SafAMD
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Retinal Function; Neuroprotection
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saffron (Active Comparator): Crocus Sativus extract
  Interventions: Dietary Supplement: Saffron
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saffron — Saffron 20 mg/day supplementation
  Arms: Saffron
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a pilot interventional study whose aim is to determine the effect of a dietary supplementation with a Crocus Sativus extract, Saffron, on macular cone-mediated function in patients with early age-related macular degeneration (AMD). Pre-clinical evidence ( Maccarone R, Di Marco S, Bisti S. Saffron supplement maintains morphology and function after exposure to damaging light in mammalian retina. Invest Ophthalmol Vis Sci. 2008 Mar;49(3):1254-61.) indicates the potential effectiveness of Saffron as a retinal neuroprotectant in animal models of retinal degenerative disorders.The macular function will be tested by visual acuity and macular cone-mediated electroretinogram (focal electroretinogram, FERG) according to a standardized technique (see citations).

DETAILED DESCRIPTION:
A group of 30 AMD patients with typical lesions (drusen and/or retinal pigment epithelial defects) and relatively preserved central retinal function and visual acuity will be enrolled. AMD patients will be randomly divided into two groups: 1. placebo group [n = 15), taking for three months an oral placebo; 2. Saffron group (n = 15), taking Saffron oral treatment (20 mg/day) for three months. After three months of placebo or Saffron supplementation, patients will be tested with standard ophthalmic examination and FERGs. Then, placebo with Saffron and vice-versa will be changed to the same patients in a cross-over design. After a further three month period of placebo or study drug supplementation, patients will undergo again a standard ophthalmic examination, and FERG. Throughout the study, both patients and experimenters will be masked as to the identity of pills (i.e. whether placebo or study drug), whose identification key number will be kept in a sealed envelope that will be opened only at the completion of the study. Therapeutic compliance will be tested by careful questioning, either at two weeks of treatment (by telephone interview) or at the end of the treatment period, as well as by pill count. Main outcome measures of the study will be FERG amplitude and phase.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 yrs
* Diagnosis of Early, non exudative AMD
* Visual acuity of 20/40 or better

Exclusion Criteria:

* Concomitant ocular or systemic disorders which may affect macular function
* Drugs that may affect macular function

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Focal Electroretinogram Amplitude and Phase | 6 months

SECONDARY OUTCOMES:
Visual Acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Falsini, M.D., Principal Investigator — Catholic University, Italy
Locations (1):
- Policlinico A. Gemelli, Institute of Ophthalmology, Rome, Italy

REFERENCES:
- [Background] Maccarone R, Di Marco S, Bisti S. Saffron supplement maintains morphology and function after exposure to damaging light in mammalian retina. Invest Ophthalmol Vis Sci. 2008 Mar;49(3):1254-61. doi: 10.1167/iovs.07-0438. PMID 18326756
- [Background] Falsini B, Piccardi M, Iarossi G, Fadda A, Merendino E, Valentini P. Influence of short-term antioxidant supplementation on macular function in age-related maculopathy: a pilot study including electrophysiologic assessment. Ophthalmology. 2003 Jan;110(1):51-60; discussion 61. doi: 10.1016/s0161-6420(02)01547-6. PMID 12511345
- [Background] Falsini B, Fadda A, Iarossi G, Piccardi M, Canu D, Minnella A, Serrao S, Scullica L. Retinal sensitivity to flicker modulation: reduced by early age-related maculopathy. Invest Ophthalmol Vis Sci. 2000 May;41(6):1498-506. PMID 10798669
- [Result] Falsini B, Piccardi M, Minnella A, Savastano C, Capoluongo E, Fadda A, Balestrazzi E, Maccarone R, Bisti S. Influence of saffron supplementation on retinal flicker sensitivity in early age-related macular degeneration. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6118-24. doi: 10.1167/iovs.09-4995. Epub 2010 Aug 4. PMID 20688744